CLINICAL TRIAL: NCT03295019
Title: Clinical Evaluation of the Efficacy of "Hyaluronan" Formulation for Dry Mouth in Sleep Apnea Patients.
Brief Title: "Hyaluronan" Formulation for Dry Mouth in Sleep Apnea Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: You First Services (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: LUA-102-16
Record Dates: First submitted 2017-09-21; First posted 2017-09-27 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Dry Mouth; Xerostomia; OSA; Sleep Apnea
MeSH Terms: conditions — Xerostomia; Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Test Oral Spray (Experimental): Subjects will be instructed to mouth spray with 0.3 ml ( 2 sprays to the mouth) of their assigned mouth spray, 2 times daily (morning and evening), using only the assigned mouth spray provided for the 4 week duration of the study.
  Interventions: Device: Test Oral Spray
- Placebo Oral Spray (Placebo Comparator): Subjects will be instructed to mouth spray with 0.3 ml ( 2 sprays to the mouth) of their placebo mouth spray, 2 times daily (morning and evening), for the 4 week duration of the study.
  Interventions: Device: Placebo Oral Spray

INTERVENTIONS:
Device: Test Oral Spray — HA formulation of FDA listed ingredients
  Arms: Test Oral Spray
Device: Placebo Oral Spray — Placebo formulation without the active ingredients
  Arms: Placebo Oral Spray

SUMMARY:
During routine clinical practice, it is observed that patients with suspected obstructive sleep apnea (OSA) often reported waking up with a dry mouth during the night or in the morning. This 9 week, cross-over group, randomized, single center, study will evaluate the efficacy of a proprietary formulation in comforting dry mouth in Sleep Apnea patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patient should be above 18 years of age.
2. Patients who have been initiated on CPAP therapy after an initial diagnosis of OSAS and have developed dry mouth or have worsening of pre-existing dry mouth condition, as an effect of CPAP therapy.
3. Ability to attend visits at the research site
4. Patient should be able to read and/or understand and sign the consent form and be willing to participate in the research study
5. Have a negative history of radiation therapy to head and neck
6. Agree to abstain from the use of any products for xerostomia other than those provided in the study.
7. Agree to comply with the conditions and schedule of the study.

Exclusion Criteria:

1. Subjects with open mouth sores at study entry.
2. Any pathology that, based on the judgement of the researcher, could negatively affect the oral mucosa and subsequent treatment for xerostomia (immune disorders, etc.)
3. Subjects who are nursing, becoming pregnant or plan to become pregnant during the study period
4. Subjects currently on medication or treatment for dry mouth/xerostomia
5. Subjects < 18 years of age
6. Hypersensitivity to any of the following ingredients- HA ,xylitol and Sodium Benzoate.
7. Subjects with soft or hard tissue tumor of the oral cavity.
8. Presence of severe gingivitis
9. Chronic disease with concomitant oral manifestations other than xerostomia
10. Subjects with conditions the investigator may feel will interfere with the condition under study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2017-08-04 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
Relief from dry mouth survey using questionnaires. | 9 weeks
  Evaluate patients' perception of efficacy of a new mouth spray compared to a placebo in reducing the symptoms of dry mouth in Sleep Apnea patients. Survey will be done by distributing diaries with daily, weekly and end of study questionnaires.

CONTACTS AND LOCATIONS:
Locations (1):
- VA WNY Healthcare System, Buffalo, New York, United States